CLINICAL TRIAL: NCT02675244
Title: Evaluating the Benefit of Concurrent Tricuspid Valve Repair During Mitral Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Canadian Institutes of Health Research (CIHR) (Other Government); German Society for Thoracic and Cardiovascular Surgery (Other); Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other)
Responsible Party: Principal Investigator, Annetine Gelijns, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 08-1078-0010; 2U01HL088942-07 (NIH)
Record Dates: First submitted 2016-01-29; First posted 2016-02-05 (Estimated); Results first posted 2023-09-21 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-05

CONDITIONS: Mild Tricuspid Regurgitation; Moderate Tricuspid Regurgitation; Tricuspid Regurgitation
Keywords: Tricuspid Valve Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MVS Alone (Active Comparator): Participants will undergo mitral valve surgery alone.
  Interventions: Procedure: MVS
- MVS + TV Annuloplasty (Active Comparator): Patients will undergo mitral valve surgery and tricuspid valve annuloplasty.
  Interventions: Procedure: TV Annuloplasty; Procedure: MVS

INTERVENTIONS:
Procedure: TV Annuloplasty — TV Annuloplasty will be performed using standard surgical techniques
  Arms: MVS + TV Annuloplasty
Procedure: MVS — MVS will be performed using standard surgical techniques

SUMMARY:
The purpose of the research is to determine whether repairing a tricuspid valve (TV) in patients with mild to moderate tricuspid regurgitation (TR), at the time of planned mitral valve surgery (MVS), would improve the heart health of those who receive it compared to those who do not.

At this point, the medical community is split in their opinion on whether surgeons should routinely repair mild to moderate TR in patients who are undergoing planned mitral valve surgery, and this study will answer this question.

DETAILED DESCRIPTION:
The tricuspid valve controls the flow of blood in your heart between the right ventricle and the right atrium. TR is a condition where the valve does not close fully when it is supposed to and blood can then leak back into the right atrium. When TR becomes severe, surgery is usually performed to correct it. The purpose of the research is to determine whether repairing a tricuspid valve in patients with mild to moderate TR, at the time of planned mitral valve surgery, would improve the heart health of those who receive it compared to those who do not. There are no new or "experimental" procedures being tested in this study: both the mitral valve procedure and the tricuspid valve repair procedure are well established surgeries and are regularly performed together in patients who have severe TR. The available evidence addressing this issue is not definite: it is based on less rigorous methods of investigation, and the results have been conflicting. The study being proposed here will use rigorous scientific methods and should result in a very high level of certainty about what surgical treatment is best for patients with your condition.

This study will enroll people scheduled for mitral valve surgery with mild to moderate tricuspid regurgitation.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing MVS for degenerative MR* with (a) Moderate TR as determined by transthoracic 2D echocardiography, or (b) Tricuspid annular dimension ≥ 40 mm (index: ≥21mm/M2 BSA) and none/trace or mild TR, determined by echocardiography.
* Age ≥ 18 years
* Able to sign Informed Consent and Release of Medical Information forms

  * "Degenerative mitral valve disease refers to a spectrum of conditions in which morphologic changes in the connective tissues of the mitral valve cause structural lesions . . ., such as chordal elongation, chordal rupture, leaflet tissue expansion, and annular dilation typically resulting in mitral regurgitation due to leaflet prolapse." This definition excludes rheumatic heart disease. (Anyanwu AC, Adams DH. (2007) Etiological classification of degenerative mitral valve disease: Barlow's disease and fibroelasticity deficiency. Semin Thorac Cardiovasc Surg; 19(2): 90-6).

Exclusion Criteria:

* Functional MR
* Evidence of sub-optimal fluid management (e.g., lack of diuretics, weight in excess of dry weight) in the opinion of the cardiology investigator
* Structural / organic TV disease
* Severe TV regurgitation as determined by preoperative transthoracic echocardiography (TTE)
* Implanted pacemaker or defibrillator, where the leads cross the TV from the right atrium into the right ventricle
* Concomitant cardiac surgery other than atrial fibrillation correction surgery (PVI, Maze, LAA closure), closure of PFO or ASD, or CABG
* Cardiogenic shock at the time of randomization
* STEMI requiring intervention within 7 days prior to randomization
* Evidence of cirrhosis or hepatic synthetic failure
* Severe, irreversible pulmonary hypertension in the judgment of the investigator
* Pregnancy at the time of randomization
* Therapy with an investigational intervention at the time of screening, or plan to enroll patient in additional investigational intervention study during participation in this trial
* Any concurrent disease with life expectancy < 2 years
* Unable or unwilling to provide informed consent
* Unable or unwilling to comply with study follow up in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2016-05-26 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annetine C. Gelijns, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Richard Weisel, MD, Study Chair — Toronto General Hospital
Locations (40):
- United States (23):
  - University of Southern California, Los Angeles, California
  - Stanford University School of Medicine, Stanford, California
  - Yale University School of Medicine - Yale-New Haven Hospital, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - University of Maryland, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - MedStar Health, Columbia, Maryland
  - University of Michigan Health Services, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Columbia University Medical Center, New York, New York
  - Stony Brook Hospital, Stony Brook, New York
  - Montefiore Einstein Heart Center, The Bronx, New York
  - Mission Hospital, Asheville, North Carolina
  - Duke University, Durham, North Carolina
  - WakeMed Clinical Research Institute, Raleigh, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Baylor Research Institute, Plano, Texas
  - University of Virginia Health Systems, Charlottesville, Virginia
  - University of Wisconsin, Madison, Wisconsin
- Canada (8):
  - University of Alberta Hospital, Edmonton, Alberta
  - London Health Sciences, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - Hôpital du Sacré-Cœur de Montréal, Montreal, Quebec
  - Institut Universitaire de Cardiologie de Quebec (Hopital Laval), Québec, Quebec
- Germany (9):
  - Universitares Herzzentrum Hamburg, Berlin, Brandenburg
  - Herzzentrum Leipzig, Berlin, Brandenburg
  - University Hospital Frankfurt, Frankfurt, Hesse-Nassau
  - University Medical Center Göttingen, Göttingen, Lower Saxony
  - University Medical Center Jena, Jena, Thuringia
  - HDZ NRW Bad Oeynhausen, Bad Oeynhausen
  - Deutsches Herzzentrum Berlin, Berlin
  - Heart Center, University of Freiburg, Freiburg im Breisgau
  - German Heart Center Munich, Munich

REFERENCES:
- [Derived] Gammie JS, Chu MWA, Falk V, Overbey JR, Moskowitz AJ, Gillinov M, Mack MJ, Voisine P, Krane M, Yerokun B, Bowdish ME, Conradi L, Bolling SF, Miller MA, Taddei-Peters WC, Jeffries NO, Parides MK, Weisel R, Jessup M, Rose EA, Mullen JC, Raymond S, Moquete EG, O'Sullivan K, Marks ME, Iribarne A, Beyersdorf F, Borger MA, Geirsson A, Bagiella E, Hung J, Gelijns AC, O'Gara PT, Ailawadi G; CTSN Investigators. Concomitant Tricuspid Repair in Patients with Degenerative Mitral Regurgitation. N Engl J Med. 2022 Jan 27;386(4):327-339. doi: 10.1056/NEJMoa2115961. Epub 2021 Nov 13. PMID 34767705

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 2016 through 2018, a total of 5208 patients were screened; 885 were eligible to participate in the trial, and 401 underwent randomization
Period: Overall Study
Arm/Group | MVS Alone | MVS + TV Annuloplasty
Started | 203 | 198
Completed | 0 | 0
Not Completed | 203 | 198
Not completed — Death | 9 | 6
Not completed — Withdrawal by Subject | 3 | 6
Not completed — Lost to Follow-up | 1 | 1
Not completed — Ongoing at 2 Years | 190 | 185

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MVS Alone | MVS + TV Annuloplasty | Total
Number analyzed (Participants) | 203 | 198 | 401
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (9.7) | 66.6 (10.7) | 67.4 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 51 | 101
  Male | 153 | 147 | 300
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 6 | 6
  Not Hispanic or Latino | 192 | 187 | 379
  Unknown or Not Reported | 11 | 5 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 7 | 3 | 10
  White | 184 | 182 | 366
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 9 | 15
Region of Enrollment [Number; unit: participants]
  Canada | 43 | 44 | 87
  United States | 116 | 120 | 236
  Germany | 44 | 34 | 78
Tricuspid-valve annulus dimension (mm) [Mean (Standard Deviation); unit: mm] | 42.2 (4.7) | 42.0 (4.6) | 42.1 (4.6)
Tricuspid Regurgitation [Count of Participants; unit: Participants]
  Moderate | 76 | 73 | 149
  < Moderate | 126 | 124 | 250
  Unable to assess | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Failure
Description: The primary outcome of this trial is treatment failure defined as the composite of (1) death from any cause, (2) reoperation for TR, (3) presence of severe TR at two years post randomization or, for patients enrolled with less than moderate TR and annular dilatation, progression by two grades (i.e., from none/trace TR to moderate TR) at two years post randomization.
Time Frame: 24 Months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MVS Alone | MVS + TV Annuloplasty
Number analyzed (Participants) | 203 | 198
percentage of participants | 10.2 [6.0 to 14.5] | 3.9 [1.1 to 6.7]

2. Secondary Outcome: Number of Participants With Major Adverse Cardiac and Cerebrovascular Events (MACCE)
Description: Major Adverse Cardiac and Cerebrovascular Events (MACCE) is defined as a non-weighted composite score comprised of the following components: Death, Stroke, and Serious heart failure events
Time Frame: up to 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | MVS Alone | MVS + TV Annuloplasty
Number analyzed (Participants) | 203 | 198
Participants | 23 | 20

3. Secondary Outcome: Number of Participants With NYHA Classification I-IV
Description: Functional status will be assessed by the New York Heart Association (NYHA) Classification scale which ranges from 1 (no physical limitations) to 4 (severe limitation of physical activity).
  1. Class I - No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  2. Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  3. Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m).Comfortable only at rest.
  4. Class IV - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
  5. No NYHA class listed or unable to determine
Time Frame: at 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | MVS Alone | MVS + TV Annuloplasty
Number analyzed (Participants) | 203 | 198
Participants
  Class I | 150 | 155
  Class II | 24 | 22
  Class III | 5 | 2
  Class IV | 0 | 0
  Died | 9 | 6
  Withdrew/LTF | 4 | 7
  Missed Assessment | 11 | 6

4. Secondary Outcome: Diuretic Use
Description: The diuretic requirements of patients will be assessed.
Time Frame: 24 Months
Population: Patients with known diuretic status at 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | MVS Alone | MVS + TV Annuloplasty
Number analyzed (Participants) | 185 | 182
Participants | 55 | 41

5. Secondary Outcome: Six Minute Walk Test
Description: The total distance, in feet, walked in six minutes
Time Frame: 24 Months
Population: Patients with observed 6MWT at 24 months
Measure: Median (Inter-Quartile Range); unit: feet
Arm/Group | MVS Alone | MVS + TV Annuloplasty
Number analyzed (Participants) | 163 | 169
feet | 1440 [1184 to 1665] | 1515 [1240 to 1706]

6. Secondary Outcome: Number of Participants With Degree of TR
Description: Degree of TR assessed by echocardiography, categorized according to American Society of Echocardiography guidelines as none/mild/moderate/severe.
Time Frame: up to 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | MVS Alone | MVS + TV Annuloplasty
Number analyzed (Participants) | 203 | 198
Participants
  None/Trace | 75 | 150
  Mild | 59 | 23
  Moderate | 35 | 5
  Severe | 10 | 1
  Died | 9 | 6
  Withdrew/LTF | 4 | 7
  Missed Assessment | 11 | 6

7. Secondary Outcome: Right Ventricular Size
Time Frame: 24 Months
Reporting Status: Not Posted

8. Secondary Outcome: Number of Participants With Normal RV Function
Description: Number of Participants with Normal RV Function assessed by echocardiography.
Time Frame: up to 24 Months
Population: Patients with observed RV Function at 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | MVS Alone | MVS + TV Annuloplasty
Number analyzed (Participants) | 178 | 178
Participants | 163 | 162

9. Secondary Outcome: Peak Tricuspid Annular Velocity
Time Frame: 24 Months
Reporting Status: Not Posted

10. Secondary Outcome: Tricuspid Annular Peak Systolic Excursion (TAPSE)
Description: Degree of RV function assessed by TAPSE
Time Frame: 24 Months
Reporting Status: Not Posted

11. Secondary Outcome: Right Ventricular Fractional Area Change (RVFAC)
Description: Degree of RV function assessed by RVFAC
Time Frame: 24 Months
Reporting Status: Not Posted

12. Secondary Outcome: Pulmonary Artery Pressure
Description: Pulmonary artery pressure assessed by echocardiography.
Time Frame: up to 24 Months
Reporting Status: Not Posted

13. Secondary Outcome: Right Ventricular Volume
Description: RV Volume as measured by transthoracic 3D echocardiography.
Time Frame: 24 Months
Reporting Status: Not Posted

14. Secondary Outcome: SF-12
Description: Quality of Life assessed by SF-12. A measure of perceived health (health-related quality of life [QoL]) that describes the degree of general physical health status and mental health distress. Higher scores indicate higher levels of health. The physical and mental health scores on the 12-Item Short Form Survey (SF-12) are reported as T scores (mean, 50±10, 50 indicates the population mean with a standard deviation of 10), with higher scores indicating better health status.
Time Frame: 24 Months
Population: Patients with observed SF-12 at 24 months
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | MVS Alone | MVS + TV Annuloplasty
Number analyzed (Participants) | 181 | 183
T-Score
  Physical Health | 47.5 (10.0) | 49.1 (9.1)
  Mental Health | 54.1 (9.0) | 54.3 (8.3)

15. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire (KCCQ)
Description: Quality of Life assessed by Kansas City Cardiomyopathy Questionnaire (KCCQ). KCCQ is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life, in which higher scores reflect better health status. Scores on the Kansas City Cardiomyopathy Questionnaire (KCCQ) overall summary range from 0 to 100, with higher scores indicating a better quality of life and fewer symptoms and physical limitations associated with heart failure.
Time Frame: 24 Months
Population: Patients with observed KCCQ at 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MVS Alone | MVS + TV Annuloplasty
Number analyzed (Participants) | 184 | 185
score on a scale | 88.0 (16.5) | 90.3 (14.8)

16. Secondary Outcome: EuroQoL (EQ-5D)
Description: Quality of Life assessed by EuroQoL (EQ-5D) - a standardised instrument for use as a measure of health outcome. Scores on the EuroQol (EQ-5D) visual analogue scale range from 0 (worst imaginable health) to 100 (best imaginable health). Higher scores indicate higher levels of health.
Time Frame: 24 Months
Population: Patients with observed Euro-QOL
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MVS Alone | MVS + TV Annuloplasty
Number analyzed (Participants) | 184 | 185
score on a scale | 81.6 (15.6) | 84.0 (13.0)

17. Secondary Outcome: Survival
Description: Incidence of participants alive
Time Frame: up to 60 Months
Reporting Status: Not Posted

18. Secondary Outcome: Length of Index Hospitalization
Time Frame: average 30 days
Population: Post-surgery hospital LOS between treatment groups compared, separately by region. 1 Canadian patient in the MVS+TA group withdrew prior to discharge from the index hospitalization so do not have their LOS
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- MVS Alone - US: MVS Alone (as described previously) patients randomized in the US
- MVS + TA - US: MVS +TA (as described previously) patients randomized in the US
- MVS Alone - Canada: MVS Alone (as described previously) patients randomized in the Canada
- MVS + TA - Canada: MVS +TA (as described previously) patients randomized in the Canada
- MVS Alone - Germany: MVS Alone (as described previously) patients randomized in Germany
- MVS + TA - Germany: MVS +TA (as described previously) patients randomized in Germany
Arm/Group | MVS Alone - US | MVS + TA - US | MVS Alone - Canada | MVS + TA - Canada | MVS Alone - Germany | MVS + TA - Germany
Number analyzed (Participants) | 116 | 120 | 43 | 43 | 44 | 34
days | 6 [5 to 8] | 8 [6 to 9] | 7 [6 to 11] | 9 [7 to 14] | 11.5 [9 to 15] | 12 [9 to 16]

19. Secondary Outcome: Number of Participants With Readmission
Description: Incidence of readmissions
Time Frame: up to 24 months
Population: *2 patients in the MVS alone and 3 patients in the MVS+TA group died during the index hospitalization, 1 patient in the MVS+TA group withdrew prior to discharge from the index hospitalization - these patients are excluded from analyses of readmission by 2 years post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | MVS Alone | MVS + TV Annuloplasty
Number analyzed (Participants) | 201 | 194
Participants | 66 | 69

20. Secondary Outcome: Number of Participants With TV Reoperations
Description: Number of participants with TV reoperations
Time Frame: up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | MVS Alone | MVS + TV Annuloplasty
Number analyzed (Participants) | 203 | 198
Participants | 0 | 0

21. Secondary Outcome: Economic Measures (Inpatient Costs)
Description: Inpatient costs will be measured through the collection of hospital billing.
Time Frame: up to 60 months
Reporting Status: Not Posted

22. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: Safety as measured by frequency of serious adverse events.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | MVS Alone | MVS + TV Annuloplasty
Number analyzed (Participants) | 203 | 198
Participants | 109 | 109

23. Secondary Outcome: Gait Speed Test
Description: Frailty will be assessed using the Gait Speed Test, which measures the average speed of three 5 meter walks
Time Frame: 24 months
Population: Patients with observed gait speed test at 24 months
Measure: Median (Inter-Quartile Range); unit: m/s
Arm/Group | MVS Alone | MVS + TV Annuloplasty
Number analyzed (Participants) | 164 | 167
m/s | 1.3 [1.0 to 1.7] | 1.3 [1.1 to 1.7]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | MVS Alone | MVS + TV Annuloplasty
All-Cause Mortality (participants affected / at risk) | 9/203 | 6/198
Serious Adverse Events (participants affected / at risk) | 109/203 | 109/198
Other Adverse Events (participants affected / at risk) | 74/203 | 61/198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MVS Alone (N=203) | MVS + TV Annuloplasty (N=198)
Bleeding (Vascular disorders) | 12 (13) | 7 (8)
Cardiac Arrhythmias - Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Arrhythmias - Sustained ventricular arrhythmia requiring defibrillation or cardioversion (Cardiac disorders) | 2 (2) | 2 (2)
Cardiac Arrhythmias - Sustained supraventricular arrhythmia requiring drug treatment or cardioversio (Blood and lymphatic system disorders) | 45 (56) | 30 (38)
Cardiac Arrhythmias - Cardiac conduction abnormalities or sustained bradycardia requiring PPM (Cardiac disorders) | 5 (5) | 28 (28)
Pericardial Fluid Collection (Cardiac disorders) | 3 (3) | 3 (3)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 16 (20) | 8 (10)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Hepatic Dysfunction (Hepatobiliary disorders) | 2 (2) | 0 (0)
Major Infection - Localized (Infections and infestations) | 15 (18) | 15 (16)
Major Infection - Endocarditis (Infections and infestations) | 1 (1) | 2 (2)
Major Infection - Sepsis (Infections and infestations) | 11 (12) | 5 (5)
Myocardial Infarction (Non- Procedure Related) (Cardiac disorders) | 2 (2) | 2 (2)
Myocardial Infarction - Peri-CABG (Cardiac disorders) | 1 (1) | 0 (0)
TIA (Vascular disorders) | 1 (1) | 2 (2)
Ischemic Stroke (Vascular disorders) | 3 (3) | 9 (9)
Hemorrhagic Stroke (Nervous system disorders) | 1 (1) | 1 (1)
Toxic Metabolic Encephalopathy (Nervous system disorders) | 3 (3) | 4 (4)
Seizure (Nervous system disorders) | 2 (3) | 3 (3)
Renal Failure (Renal and urinary disorders) | 5 (5) | 3 (3)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 5 (7)
Heart Failure (Cardiac disorders) | 13 (21) | 9 (14)
Arterial Non-CNS Thromboembolism (Vascular disorders) | 2 (2) | 0 (0)
Venous Thromboembolic Event (Vascular disorders) | 2 (2) | 0 (0)
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Other SAE (General disorders) | 47 (71) | 37 (52)
Neurological Dysfunction - Other (Nervous system disorders) | 1 (1) | 0 (0) — SAE term did not meet specific CTCAE event criteria
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MVS Alone (N=203) | MVS + TV Annuloplasty (N=198)
Cardiac Arrhythmias -Sustained supraventricular arrhythmia requiring drug treatment or cardioversion (Cardiac disorders) | 57 (62) | 44 (47)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 9 (9)
Major Infection - Localized (Infections and infestations) | 19 (21) | 15 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-01-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT02675244/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/44/NCT02675244/SAP_001.pdf